CLINICAL TRIAL: NCT00374855
Title: Protocol H8D-MC-EMBH PPAR Alpha (LY518674): a Phase 2 Dose-Response Study to Evaluate the Blood Pressure-Lowering Effect in Essential Hypertension
Brief Title: A Study in People With Mild Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9593; H8D-MC-EMBH
Record Dates: First submitted 2006-09-08; First posted 2006-09-12 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2007-05

CONDITIONS: Mild Hypertension
MeSH Terms: interventions — PPAR alpha; Hydrochlorothiazide

INTERVENTIONS:
Drug: PPAR alpha
Drug: Hydrochlorothiazide
Drug: Placebo

SUMMARY:
The primary objective of this study is to test the hypothesis that LY518674, administered for 6 weeks to patients with mild hypertension, reduces Systolic Blood Pressure, compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Are men and women between 18 and 70 years of age, inclusive
2. Have given signed informed consent to participate in this study
3. Are diagnosed with mild essential hypertension at screening (currently untreated or treated with monotherapy)

Exclusion Criteria:

1. Secondary or malignant hypertension
2. Have or have had a history of hyperlipidemia within 3 months of screening requiring treatment
3. Any previous cardiovascular disease other than hypertension
4. Type 1 or 2 diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153
Dates: Start 2006-09; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that LY518674, administered for 6 weeks to patients with mild hypertension, reduces 24-hour mean ambulatory Systolic Blood Pressure, compared with placebo.

SECONDARY OUTCOMES:
Determine the duration and consistency of the reduction in BP over the course of a day, relative to placebo, after 6 weeks of treatment with LY518674 when taken once daily
Evaluate the population dose and exposure response relationships of LY518674 for lowering the mean SBP and DBP during the 24 hour period, using ABPM during a 6 week treatment period
Evaluate the population dose, exposure, and time response relationships of LY518674 for lowering the mean SBP and DBP during the 8 hour awake period, using ABPM during a 6 week treatment and following cessation of dosing
Compare the effect of LY518674 on CBPM SBP and DBP with that of placebo
Determine the percentage of responders to LY518674, relative to placebo, as defined by patients who achieve target BP goals of CBPM SBP <140 mm Hg and/or DBP 90 mm Hg, or a CBPM SBP decrease of at least 10 mm Hg
Evaluate the effects of LY518674, relative to placebo, on plasma levels of total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), HDL-C, triglycerides (TG), and high-sensitivity C-reactive protein (hsCRP)
Evaluate the safety and tolerability effects of LY518674, relative to placebo, in patients with mild hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (10):
- Sweden (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Åmål
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Falköping
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Gothenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Järfälla
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Luleå
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Mönsterås
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Rättvik
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Skellefteå
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Stockholm

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com